CLINICAL TRIAL: NCT06644248
Title: Development and Evaluation of an Artificial Intelligence Model for Cervical Cancer Detection From Colposcopic Images
Brief Title: AI Model for Cervical Cancer Detection From Colposcopy Images
Status: Recruiting | Type: Observational
Sponsor: Bangladesh University of Engineering and Technology (Other)
Responsible Party: Principal Investigator, Taufiq Hasan, PhD, Associate Professor, Bangladesh University of Engineering and Technology
Other Study IDs: ISMC/Admin/2023/2149
Record Dates: First submitted 2024-07-30; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Cancer; Colposcopy; Deep Learning; Transformation Zones
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Self reported uterine distress undergoing colposcopic evaluation: The study group consists of women undergoing cervical cancer screening. This includes those with suspected cervical abnormalities identified through initial cytology or HPV tests and referred for colposcopy. The study group also includes women without apparent cervical abnormalities to ensure a comprehensive dataset. The aim is to develop an AI model capable of accurately diagnosing cervical cancer and identifying transformation zones in colposcopic images. This diverse group allows for the evaluation of the AI model across a wide range of conditions and exposures, enhancing its generalizability and clinical utility.
  Interventions: Diagnostic Test: Colposcopy

INTERVENTIONS:
Diagnostic Test: Colposcopy — The intervention involves the use of colposcopy, a diagnostic procedure to visually examine the cervix using a colposcope. The procedure includes the application of saline, acetic acid, and iodine solutions to enhance the visualization of cervical tissues and identify abnormalities. The dosage form includes applying these solutions directly to the cervical area. The frequency of the intervention is typically a single session per patient, with the duration of the procedure lasting approximately 10-15 minutes. This study aims to utilize an AI model to analyze the colposcopic images obtained during the procedure to improve the accuracy and efficiency of cervical cancer detection.

SUMMARY:
Cervical cancer is a significant health issue, particularly in low-income countries, where late diagnosis and limited access to screenings contribute to high mortality rates. This study aims to develop and evaluate an artificial intelligence (AI) model to analyze colposcopic images for detecting cervical cancer more accurately and efficiently. Colposcopy, a procedure used to examine the cervix for signs of cancer, relies heavily on doctors' expertise, leading to inconsistent results. The current gold standard, colposcopy-directed biopsy, is invasive and can cause complications. The hypothesis is that an AI model can outperform traditional methods in identifying cervical abnormalities, providing a reliable and scalable solution for early detection, especially in underserved areas. By automating the analysis process, the AI model aims to reduce reliance on trained personnel, making cervical cancer screening more accessible and improving early diagnosis and treatment outcomes. The study will create a diverse dataset of colposcopy images from various sources and develop the AI model. The model's performance will be validated in clinical settings, assessing its accuracy in classifying cancer stages and identifying transformation zones. The impact on early detection, patient outcomes, and model usability will be evaluated, as well as its generalizability across different healthcare environments. The goal is to enhance the accuracy and efficiency of cervical cancer screening, ultimately reducing mortality rates and improving patient care.

DETAILED DESCRIPTION:
The study aims to develop an AI model to improve cervical cancer screening by analyzing colposcopic images. The study is a prospective and retrospective case-control study conducted at Ibn Sina Medical College Hospital in Dhaka, Bangladesh. The primary goal is to leverage deep learning techniques to enhance the accuracy and efficiency of cervical cancer detection, particularly in low-resource settings. Cervical cancer remains a significant health challenge, particularly in low- and middle-income countries where access to timely screening and treatment is limited. Colposcopy is a diagnostic procedure used to examine the cervix for signs of disease. Traditional colposcopy is highly dependent on the clinician's experience, leading to subjectivity and potential inaccuracies. This research proposes using AI to automate the analysis of colposcopic images, aiming to provide a more objective and reliable diagnostic tool. The primary objectives are to curate a comprehensive dataset of colposcopy images and develop an AI model capable of accurately classifying transformation zones and detecting cervical abnormalities. Specific objectives include clinical validation of the AI model's performance, assessing the model's usability in clinical workflows, evaluating the impact of the AI model on early detection of cervical cancer, ensuring the model's generalizability across diverse datasets, and investigating the model's effectiveness as a clinical decision support tool. Inaccuracies in traditional vision screening and a shortage of trained personnel in low-resource settings hinder effective cervical cancer screening. The AI model aims to mitigate these issues by providing an automated, scalable, and cost-effective solution. By improving the accuracy and accessibility of cervical cancer screening, this research has the potential to significantly impact patient outcomes in resource-limited environments. The study involves both prospective and retrospective data collection. Colposcopic images and relevant clinical metadata will be gathered from patients at the study sites. The data will be used to train and validate the AI model. Inclusion criteria for the study are women aged 18 or older who are willing to participate in cervical cancer screening and have no history of hysterectomy. Exclusion criteria include pregnant women and individuals with severe medical conditions that could affect screening results. The target population includes confirmed cervical cancer patients and individuals with suspected cervical abnormalities. Data from individuals with normal cervical conditions will also be included to facilitate unsupervised learning. Sample size calculations will follow established methodologies for evaluating diagnostic performance, considering factors such as sensitivity, specificity, and disease prevalence. The study includes several quality assurance measures to ensure data accuracy and reliability. A quality assurance plan addresses data validation and registry procedures, including site monitoring and auditing. Data checks will compare registry entries against predefined rules for range and consistency. Source data verification will be conducted by comparing registry data with external sources such as medical records. Standard Operating Procedures (SOPs) will cover registry operations, including patient recruitment, data collection, data management, data analysis, adverse event reporting, and change management. Sample size assessment specifies the number of participants required to demonstrate the model's effectiveness. A plan for addressing missing data includes strategies for handling unavailable or inconsistent data. The statistical analysis plan outlines the methods for evaluating the AI model's performance, including sensitivity, specificity, and accuracy metrics. The analysis will also consider the model's generalizability across different datasets and its impact on clinical decision-making and patient outcomes. This research seeks to develop an AI-based solution to improve cervical cancer screening accuracy and accessibility, particularly in low-resource settings. By addressing the limitations of traditional colposcopy and leveraging advanced computational techniques, the study aims to provide a scalable and effective tool for early detection of cervical cancer, ultimately improving patient outcomes and reducing mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of age 18 years or older can be selectedas subjects.
* Individuals willing to participate in cervical cancerscreening.
* Availability for colposcopic examination.
* Women with no history of hysterectomy (total removalof the uterus).
* Women with no current or prior diagnosis of cervicalcancer.
* Availability of relevant medical records forconfirmation and comparison purposes.

Exclusion Criteria:

* Pregnant women, given the potential impact onscreening results and the need for specialconsiderations during pregnancy.
* Individuals with severe medical conditions orcircumstances that may make colposcopic examinationinappropriate or unsafe.
* Patients with conditions that could interfere with theaccuracy of the screening results, such as severevaginal bleeding.
* Follow-up screenings.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The eligibility for this clinical study is based on gender, specifically targeting female participants. This criterion is due to the study's focus on cervical cancer, a condition that exclusively affects individuals with a cervix. Participants must be women who are referred for colposcopy due to abnormal cytology or HPV test results. The inclusion of only female participants ensures that the study accurately addresses the detection and diagnosis of cervical cancer through colposcopic examination and the evaluation of the AI model's performance in this context. No male participants are included as cervical cancer does not occur in the male population.
Study Population: The study cohort will consist of women referred to colposcopy clinics due to abnormal cytology, positive HPV tests, or self-reported cervical distress requiring evaluation. Participants will be sourced from listed primary care clinics, ensuring a diverse sample across age groups and socioeconomic backgrounds for comprehensive representation. The project aims to assess the AI model's efficacy in detecting cervical anomalies in a real-world clinical context, evaluating its performance across diverse populations and addressing the unique challenges of cervical cancer screening in varied healthcare settings.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2025-02-11 (Estimated)

PRIMARY OUTCOMES:
Swede Score Evaluation | 12 hours
  The Swede score will be used to evaluate the severity of cervical abnormalities identified in colposcopic images. This scoring system assesses various colposcopic findings, including acetowhiteness, lesion size, and vascular patterns, to determine the effectiveness of the AI model in evaluating cervical abnormalities.

SECONDARY OUTCOMES:
Transformation Zone Classification Accuracy | 12 hours
  The metric used includes accuracy, precision, recall, and F1-score for the classification of the transformation zone (TZ) in colposcopic images by the AI model. These metrics will assess the effectiveness of the AI model in identifying and classifying the transformation zone in colposcopic images.

CONTACTS AND LOCATIONS:
Overall Officials: Taufiq Hasan, Taufiq, Principal Investigator — Department of Biomedical Engineering, BUET, Dhaka - 1205.
Locations (1):
- Ibn Sina Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT06644248/Prot_SAP_ICF_000.pdf